CLINICAL TRIAL: NCT07095673
Title: Person-Centered Approach to Promoting Healthy Weight and Reducing Pain in Older Adults in Camden-New Jersey
Brief Title: HealthyWE: Achieving a Healthy Weight and Reducing Pain
Acronym: HealthyWE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Thomas A. Dahan, Ph.D., Assistant Teaching Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro2022001911
Record Dates: First submitted 2025-07-09; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Obesity &Amp; Overweight
Keywords: obesity reduction; self-efficacy; exercise intervention; low-income community; integrative strategies
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy WE (Other): Sixty (60) adults residing in the Housing Authority of the City of Camden will be recruited to be engaged in HealthyWE program to be completed in 4 weekly coaching sessions. Treatment adherence refers to the extent to which interventions are delivered as prescribed
  Interventions: Behavioral: HealthyWE

INTERVENTIONS:
Behavioral: HealthyWE — Following baseline assessment, 60 residents will be enrolled in HealthyWE Corps program. HealthyWE Corps includes training sessions on keeping a healthy weight, healthy diet, and mental health wellness. The content of the HealthyWE protocol was carefully designed choosing skills shown to be efficacious in keeping a healthy weight and reducing pain. Self-efficacy theory guides the intervention. Behavioral interventions for reducing and managing obesity focus on building adults' self-management skills to be implemented in their daily lives. To achieve the therapeutic effects, individuals have to execute self-management skills in their daily lives. Self-efficacy is defined as a person's belief in his/her ability to perform specific skills to reduce and manage obesity.

SUMMARY:
The goal of this project was to reduce and manage obesity and increase self-efficacy for keeping a healthy weight and improve pain, quality of life, and mental health symptoms among 60 adults aged 19 and older in Camden City, New Jersey. The City of Camden has an adult obesity rate of 44.1%. Obesity and aging are significant contributing factors to increased utilizations of healthcare services. Obesity is a major risk factor for non-communicable illnesses such as cardiovascular disease, type 2 diabetes, hypertension, dyslipidemia, pain, and mental health. Physical activity is effective in reducing and managing obesity. However, personal barriers (e.g., lack of time for physical activity, physical capability to perform physical activities, competing demands), built environment (e.g., safe spaces for physical activities), climate changes (e.g., heat waves and extreme weather which prevent outdoor physical activities), and systematic barriers (e.g., intervention availability) hamper obesity prevention and management in older adult population. To help older adults keep a healthy weight, our team has adapted and delivered the effective person-centered integrative interventions: HealthyWE: Keeping a Healthy Weight program to older adults in Camden New Jersey. Completion of the project will build a strong community capacity in Camden to sustain a community effort to reduce obesity and pain.

DETAILED DESCRIPTION:
The purpose of this project was to pilot test a web-based weight loss program called HealthyWE will help adults lose weight and decrease pain among adults in Camden City New Jersey. The proposed study was a one group pretest and posttest design.

A. Aims

1. Between 10/1/2023 and 9/30/2024, Rutgers University overarching goal was to reduce obesity incidence from 45% to 32% (30% reduction based on Camden County Health Department data for adult obesity) among adults living in Camden City and increase self-efficacy for keeping a healthy weight to improve quality of life and mental health symptoms.
2. Between 10/1/2023 and 5/1/2024, Rutgers University sought to recruit 60 overweight and obese participants into the HealthyWE Corps, an obesity reduction/prevention program focused on educating the public about nutrition, exercise, and a healthy mind at three sites in the city of Camden.
3. Between 10/1/2023 and 10/1/2024, Rutgers University hired and managed 3 instructors (one each in the areas of community-based nutrition education, exercise and physical activity, and mental health wellness) to lead HealthyWE Corps participants through lessons and activities focused on these areas between 1/16/2024 and 5/1/2024. Activities are designed to increase HealthyWE Corps participants capacity to engage other community members in activities related to these focus areas.
4. Between 5/1/2023 and 9/30/2024, Rutgers University assessed feasibility of HealthyWE Corps by examining (a) program accrual of adults (N=60 by 1/16/2024); (b) protocol adherence (>80% adherence to protocol, which involves the degree to which program participants engage in program activities between 5/1/2023 and 9/30/2024); and (c) participant retention (>80% data collected at evaluation appointments: pre-assessment, mid-point assessment, post-assessment).
5. Between 5/1/2024 and 9/30/2024, Rutgers University evaluated the self-efficacy for keeping a healthy weight and program adherence with expected outcome of 50% of HealthyWE Corps participants demonstrating good to excellent self-efficacy and program adherence through daily use of a FitBit-style tracker device to record their daily exercise and other health information (no health information will be collected for research purposes from the tracker device).
6. Between 5/1/2024 and 9/30/2024, Rutgers University conducted program outcome evaluation on 60 HealthyWE Corps participants to assess the effectiveness of the HealthyWE Corps program on primary outcomes of weight, BMI, and self-efficacy, and secondary outcomes of quality of life and mental health symptoms and participants overall satisfaction with the program.

1.2 Research Significance Obesity remains a major public health crisis. According to the Centers for Disease Control and Prevention, the prevalence of obesity is higher among adults (41.5%) than younger adults (39.5%). With respect to race and ethnicity, the overall prevalence of obesity is higher among non-Hispanic Black (49.9%) and Hispanic adults (45.6%) than among non-Hispanic White (41.4%). African American women have the highest prevalence of obesity (54.8%), followed by Hispanic women (50.6%) and Hispanic men (43.1%), respectively. Severe obesity is more prevalent among women, Black Americans, and low-income adults. The public health impact of obesity is profound. It is a major risk factor for non-communicable illnesses such as cardiovascular disease, type 2 diabetes, hypertension, dyslipidemia, pain, and mental health. Obesity increases risk for pain and worsens overall pain severity and interference. Further, individuals with obesity report poor physical and psychological quality of life and disproportionately reduces life expectancy. Obesity and aging are significant contributing factors to increased utilizations of healthcare services.

Camden City in New Jersey is at high risk for poorer health outcomes (e.g., obesity, pain) for a myriad of socio-economic factors and a lack of a built environment that supports health. Camden City in New Jersey is ranked as Number Four top overweight cities in the United States with 44.1% of the adult population are obese and 44.6% of the adults do not engage in leisure time activity.9 The disparate rate of obesity occurring in Camden residents is the result of complex interaction of social determinants of health (e.g., poverty, education, and housing) and neighborhood structural barriers. Camden City in New Jersey represents many overburdened communities in the United States where minority or low-income communities bear disproportionately poor human health outcomes (e.g. obesity) and environmental risks. The 8.9-mile city is the home to 73,236 residents with the average household income of $41,180 and the poverty rate of 36%. The predominant races of the residents are Black (41.4%), Hispanic (27.6%), and White (23.5%).

As a complex disease, obesity is the accumulation of body fat and an inflammatory condition that results from many contributing factors, such as malnutrition, lack of physical activity, stress, and inadequate sleep.18-22 The standard criterion to define obesity is a body mass index (BMI) 30 kg/m2 or higher. Individuals who are obese are typically on the receiving end of health education and behavioral change recommendations to increase their intake of fresh fruits and vegetables along with prescriptions for physical activity of 30 minutes a day for most days of the week. In Camden, however, these recommendations are hampered by a lack of access to safe spaces for physical activity and healthy food. In addition, personal barriers (e.g., lack of time for physical activity, physical capability to perform physical activities, competing demands, cost of healthy food, built environment (e.g., safe spaces for physical activities), climate changes (e.g., heat waves and extreme weather which prevent outdoor physical activities), and systematic barriers (e.g., intervention availability) further hamper obesity prevention and management. Prevention and management of obesity necessitates integrative approach in communities like Camden to take into considerations of individual's physical capacity, built environment for physical activity and access to good nutrition.

Rutgers University has a well-earned international reputation for excellence that is integral to our priority of addressing healthcare disparities both in the U.S. and globally. Rutgers University-Camden has been named a Minority Serving Institution (MSI) by the Department of Education under Titles III and V of the Higher Education Act. Advancing health equity is the highest priority of Rutgers School of Nursing-Camden. Social justice is the fundamental value and unifying theme informing our School of Nursing strategic direction. Faculty and students believe a person's zip code should not determine the quality of their health care. However, we recognize neighborhoods and built environments do in fact make an enormous impact on access to care, good health, and well-being. The zip codes for the project are 08104 and 08105 in the City of Camden.

Based on the Centers for Disease Control and Prevention recommendations for prevention and management of overweight and obesity and personal and structural barriers faced by low-income older adult residents in Camden City, our team has adapted the effective and person-centered integrative interventions: HealthyWE Corps. This program is an AmeriCorps service program adapted to increase participant knowledge of and engagement in healthy nutrition, healthy exercise, and mental health wellness. Community service has been demonstrated to be an effective method of increasing individual self-efficacy and evidence for being effective for reducing weight in adults.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 19
* BMI of > 25

Exclusion Criteria:

* Adults with BMI of less than 25
* Adults who are not active:
* with activity participation limitations
* with disability (physical, mental)
* impairment (vision, hearing and memory loss, cognitive)
* dementia
* Alzheimer's disease (AD).

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index | 3 intervals: baseline, 6-week follow up and 14-week follow up.
  A stand-on bioimpedance analysis (BIA) device (InBody 520, Biospace Co., Ltd., Cerritos, CA, USA) is used to automatically calculate BMI (kilogram/meters squared, kg/m2). Obesity is defined as a BMI>30 kg/m2. The Inbody 520 multifrequency BIA device is also used to measure body fat percentage, and body fat mass using impedance at 5, 50, and 500 kHz.

SECONDARY OUTCOMES:
Pain Severity and Interference | 3 intervals: baseline, 6-week follow up and 14-week follow up.
  Pain severity and pain interference are measured using the Brief Pain Inventory-Short Form (BPI-SF).40 The BPI-SF consists of four items assessing pain severity (worst, least, average, and current pain) and seven items assessing pain interference in the past week. The BPI-SF uses an 11-point response scale, with options ranging from 0 (no pain or no interference) to 10 (pain as bad as you can imagine or completely interferes). Separate composite scores are computed for pain severity and pain interference by averaging items, with high scores indicating greater pain severity and pain interference. The BPI-SF has demonstrated good reliability and validity.40-41
Quality of Life (PROMIS GHS) | baseline, 6-week follow up and 14-week follow up.
  The 10-item V1.2 Patient Reported Outcome Measure Information System Global Health Scale (PROMIS GHS), (a= 0.80-0.86)42 that captures self-perception of quality of life in terms of mental and physical health, social connection, emotional state, pain and fatigue on a scale from 1 (poor), 2 (fair), 3 (good), 4 (very good) to 5 (excellent).
Mental Health Symptoms | baseline, 6-week follow up and 14-week follow up.
  The 2-item Patient Health Questionnaire (PHQ-2) screen tool with a reported sensitivity=100% (specificity=77%, AUC=0.88) will be used to assess depression;43-44

OTHER OUTCOMES:
Self-efficacy for Achieving a Healthy Weight | baseline, 6-week follow up and 14-week follow up.
  This will be assessed using an adapted subscale of Self-Efficacy Scale.39 This subscale contains fifteen items that assess adults' certainty about their degree of performing home-based muscle-tightening breathing and pumping exercises, nutrition-balanced and portion-appropriate diet, hydration, large muscle exercises, and sleep. The items are answered on a 10 (very uncertain) to 100 (very certain) scale and averaged to obtain an overall score. This measure is a primary indicator of program adherence and should predict improved program outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Dahan, PhD, Principal Investigator — Rutgers, the State University of NJ
Locations (1):
- School of Nursing Camden, Camden, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Immediately following publication with no end data.
Access Criteria: Anyone who wishes to access the data for any purpose.